CLINICAL TRIAL: NCT02634710
Title: Pilot Study Evaluating Hypofractionated Pre-operative Radiation Therapy for Soft Tissue Sarcomas of the Extremity and Chest-wall
Brief Title: Hypofractionated Pre-operative Radiation Therapy for Soft Tissue Sarcomas of the Extremity and Chest-wall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Ciani M Ellison, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25722
Record Dates: First submitted 2015-11-04; First posted 2015-12-18 (Estimated); Results first posted 2023-06-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypofractionated Radiation Therapy (Experimental): Radiation treatment in which the total dose of radiation is divided into large doses and treatments are given every other day. Hypofractionated radiation therapy is given over a shorter period of time (fewer days or weeks) than standard radiation therapy.
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Treatments will have a minimum of a 48-hour interfraction interval. Treatments will be completed over 20 days maximum.

SUMMARY:
This is a nonrandomized Phase II pilot protocol to determine the feasibility, toxicity and disease control (local control, overall and progression-free survival) using hypofractionated preoperative radiation therapy in patients with primary localized soft tissue sarcomas (STS).

DETAILED DESCRIPTION:
BACKGROUND OVERVIEW: Hypofractionation has several potential advantages over conventional radiation. First, the biological equivalent dose to the tumor is higher with hypofractionation than it is with conventional radiation. In between radiation treatments there is repair of the radiation damaged cancer cells (on a cell survival curve this region of repair is referred to as the "shoulder" of the curve). Some cell lines are better at repair than others. Sarcoma is often referred to as a "radioresistant" tumor, which means that sarcoma cell lines have a larger capacity for radiation repair than do other cell lines. A treatment that can deliver a high dose in fewer fractions can potentially overcome some of this repair. There is a concept in radiation known as "biologically equivalent dose" (BED) which states that a higher dose per fraction results in more tumor kill than a lower dose per fraction. For example, radiation delivered to a total of 60 Gy in three 20 Gy fractions is the equivalent of 150 Gy in 2 Gy fractions.

BACKGROUND RATIONALE: It is important to conduct this study because hypofractionation not only decreases treatment package time and cost of care, but it also potentially improves patient convenience and quality of life and could impact radiologic and pathologic variables in a positive way by leading to more tumor cell kill. This could potentially change the paradigm of the current management of STS of the extremity and chest-wall.

HYPOTHESIS: Preoperative hypofractionated radiation therapy for localized soft tissue sarcomas (STS) will result in local control and toxicity similar to conventional fractionation with less cost, more patient convenience and decreased overall treatment time.

TREATMENT: Image-guided radiation therapy is mandatory. PREOPERATIVE: (1) Either 3D conformal radiotherapy or intensity modulated radiation therapy (IMRT). (2) A prescription dose of 35 Gy in 5 fractions given every other day with at least 48 hours in between each fraction will be prescribed to cover 95% of the planning target volume. TREATMENT SCHEDULE: Treatments will have a minimum of a 48-hour interfraction interval. Treatments will be completed over 20 days maximum.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Core needle biopsy obtained
* Pathologic confirmation of primary soft tissue sarcoma of the upper or lower extremity or chest-wall.
* Stage I-III Soft Tissue Sarcoma of the extremity without evidence of metastatic disease
* Medically operable
* No prior radiotherapy to primary site or adjacent site that results in overlapping radiation fields.
* MRI obtained of the affected extremity or chest-wall
* CT chest acquired to assess distant disease
* Karnofsky Performance Status (KPS) 60 or above
* Informed consent obtained prior to study entry

Exclusion Criteria:

* Patients who have metastatic disease
* Pregnant women
* Women of childbearing potential and male participants must practice adequate contraception.
* Disease pathology other than sarcoma subtypes
* Patients with a history of metastatic disease from a primary other than sarcoma
* Patients who cannot undergo MRI as part of pre-treatment or treatment planning process
* STS of non-extremity or chest-wall regions
* Tumor size ≥ 20 cm maximal dimension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciani Ellison, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bedi M, Singh R, Charlson JA, Kelly T, Johnstone C, Wooldridge A, Hackbarth DA, Moore N, Neilson JC, King DM. Is 5 the New 25? Long-Term Oncologic Outcomes From a Phase II, Prospective, 5-Fraction Preoperative Radiation Therapy Trial in Patients With Localized Soft Tissue Sarcoma. Adv Radiat Oncol. 2022 Jan 25;7(3):100850. doi: 10.1016/j.adro.2021.100850. eCollection 2022 May-Jun. PMID 35647402

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypofractionated Radiation Therapy
Started | 35
Completed | 31
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Local Disease Control Assessed by Physical Examination
Description: This measure will capture the number of subjects experiencing a recurrence of the primary lesion assessed by physical examination.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
Participants | 0

2. Primary Outcome: Local Disease Control Assessed by Magnetic Resonance Imaging (MRI)
Description: This measure is the number of subjects experiencing a recurrence of the primary lesion as assessed by MRI.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
Participants | 0

3. Secondary Outcome: Musculoskeletal Tumor Rating Scale (MSTS) Score
Description: Toxicity will be assessed at specific times the Musculoskeletal Tumor Rating Scale. The MSTS evaluates: pain, function, emotional acceptance, hand positioning, dexterity and lifting ability, using a six-item Likert scale ranging from 0 (worst condition) to 5 (best condition). The individual scores are added for the MSTS Score, range 0 to 30. A higher score indicates better function.
Time Frame: Baseline, prior to surgery and 24 months after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
units on a scale
  Baseline | 29 (1.05)
  Prior to Surgery | 28.3 (2.06)
  2 years | 27.3 (2.47)

4. Secondary Outcome: Disease-free Survival
Description: Disease-free survival will measure the time in months from initiation of radiation therapy until documented recurrence of disease. Patients who are disease-free and alive at the time of analysis will be censored at the time of their last follow-up. Patients will be assessed for disease-free survival at 2 years.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
Participants | 32

5. Secondary Outcome: Overall Survival
Description: Overall survival will measure the time from initiation of radiation therapy until documented death from any cause. Patients who are alive at the time of analysis will be censored at the time of their last follow-up. Patients will be assessed for overall survival at 2 years.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
Participants | 32

6. Secondary Outcome: Radiologic Changes Due to Hypofractionated Radiation.
Description: This measure will assess the size of enhancement due to hypofractionated radiation.
Time Frame: 4 weeks after radiation therapy
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
cubic centimeters | -16.2 (25)

7. Secondary Outcome: Pathologic Changes Due to Hypofractionated Radiation.
Description: This measure will capture the fibrosis present in tissue specimens as a percent.
Time Frame: 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: percentage of tumor specimen
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
percentage of tumor specimen
  Necrosis | 17.5 (26.4429)
  Fibrosis | 20 (32.5364)
  Viable Cells | 50 (31.9287)

8. Secondary Outcome: Treatment-related Necrosis and Fibrosis
Description: Number of participants who experienced treatment-related necrosis and fibrosis ≥90%.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 35
Participants
  Treatment-related necrosis | 4
  Treatment-related fibrosis | 4

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Hypofractionated Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 4/35
Serious Adverse Events (participants affected / at risk) | 19/35
Other Adverse Events (participants affected / at risk) | 20/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated Radiation Therapy (N=35)
Cardiac arrest (Cardiac disorders) | 1 (1)
Hyper parathyroidism (Endocrine disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Wound infection (Infections and infestations) | 3 (3)
Wound infection (Infections and infestations) | 4 (4)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated Radiation Therapy (N=35)
Edema limbs (General disorders) | 3 (3)
Localized edema (General disorders) | 3 (3)
Radiation dermatitis (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT02634710/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT02634710/ICF_001.pdf